CLINICAL TRIAL: NCT03611127
Title: The Impact of Early Pulmonary Rehabilitation on the Multidimensional Aspects of Dyspnea and Exercise Performance Following Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: The Impact of Early Pulmonary Rehabilitation on Multidimensional Aspect of Dyspnea in COPD Patients After Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Shoukri, Associate Professor of Pulmonary medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR_15_11404_SHOUKRI
Record Dates: First submitted 2018-07-10; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early pulmonary rehabilitation (EPR) (Experimental): early pulmonary rehabilitation started shortly after hospital discharge for COPD exacerbation.
  Interventions: Other: pulmonary rehabilitation
- Usual care (UC) (No Intervention): No pulmonary rehabilitation for this group

INTERVENTIONS:
Other: pulmonary rehabilitation — pulmonary rehabilitation standardized program
  Arms: early pulmonary rehabilitation (EPR)

SUMMARY:
Acute exacerbations of chronic obstructive pulmonary disease (AECOPD) are associated with severe dyspnea and exercise intolerance. Early pulmonary rehabilitation (EPR) may lead to improvements in dyspnea and exercise tolerance, as it does in stable COPD patients.

DETAILED DESCRIPTION:
One hundred and six patients admitted in a university hospital with AECOPD were randomized after discharge to either EPR for 8 weeks (EPR group) or usual care (UC) (UC group). All patients carried out the following initially and after 8 weeks: spirometry, 6minute walk test (SMWT), and a symptom-limited incremental cycle cardiopulmonary exercise test (CPET), and different dyspnea dimensions evaluation as following: Dyspnea intensity during incremental exercise using Borg scale, dyspnea 12 questionnaire and COPD assessment test (CAT) to assess sensory perceptual, affective distress, and symptom impact domains respectively.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized COPD patients with a diagnosis of AECOPD with no clinically significant arterial hypoxemia at rest or on exercise (resting percutaneous oxygen saturation (SpO2) > 90% or a sustained decrease of < 4% during exercise) were recruited. Diagnosis of COPD, AECOPD and spirometric assessment of airflow limitation severity was based on Global Initiative for Chronic Obstructive Lung Disease (GOLD)

Exclusion Criteria:

* Patients with a prior diagnosis of other cardiorespiratory conditions (i.e., bronchial asthma, interstitial lung diseases, primary pulmonary hypertension, chronic congestive heart failure), as well as other conditions such as orthopedic, muscular and peripheral vascular diseases that could cause or contribute to breathlessness and exercise intolerance and/or could interfere with carrying out of exercise testing, were excluded.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
change in different aspects of dyspnea (dyspnea 12 questionnaire: scale range 0-36, with high score indicating worse dyspnea, and COPD assessment test: scale range 0-40, high score indicating worse dyspnea). | 8 weeks
  dyspnea questionnaires
change in exercise performance (borg scale during incremental exercise measuring the perceived dyspnea: scale 0-10, higher score indicating worse performance | 8 weeks
  cardiopulmonary exercise tests
change in exercise performance (test duration: longer duration measured in seconds indicating better performance) | 8 weeks
  cardiopulmonary exercise tests
change in exercise performance (Peak oxygen consumption: Higher values indicating better performance) | 8 weeks
  cardiopulmonary exercise tests

IPD SHARING:
Plan to Share IPD: No